CLINICAL TRIAL: NCT04382014
Title: Pharmacokinetic Study on Three Formulations of Curcumin With Different Carriers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MaxSimil + curcumin
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Healthy
MeSH Terms: interventions — Curcumin; Rice Bran Oil

STUDY DESIGN:
Intervention Model Description: Double-blind controlled-randomized pharmacokinetic (PK) study with crossover design (15 men and 15 women), with a minimum of 6 days between treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the research nurse will know the administration order of the different treatments administered. All plasma samples collected during the research project will be anonymized. Also, it will not be possible to identify the participant by his name since a number will be assigned to him. The code key linking the participant's name to his number will be stored, with access restricted to those designated by the principal investigator. The data file is also protected by a password.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAG fish oil + Curcumin (Experimental): The participant will arrive fasted at he research center. After installing a catheter and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of 1,5 g MAG fish oil + 400 mg curcumin. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of curcumin in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: MAG fish oil + Curcumin OR Rice bran oil + Curcumin OR Curcumin extract
- Rice bran oil + Curcumin (Active Comparator): The participant will arrive fasted at he research center. After installing a catheter and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of rice bran oil + 400 mg curcumin. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of curcumin in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: MAG fish oil + Curcumin OR Rice bran oil + Curcumin OR Curcumin extract
- Curcumin extract (Active Comparator): The participant will arrive fasted at he research center. After installing a catheter and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive 1 dose of 400 mg curcumin. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of curcumin in the plasma and a side effect questionnaire will be administered to monitor side effects.
  Interventions: Dietary Supplement: MAG fish oil + Curcumin OR Rice bran oil + Curcumin OR Curcumin extract

INTERVENTIONS:
Dietary Supplement: MAG fish oil + Curcumin OR Rice bran oil + Curcumin OR Curcumin extract — The intervention is a randomized double blind cross over design testing the pharmacokinetics of 1) curcumin combined with MAG fish oil as a carrier, 2) curcumin combined with rice bran oil as a carrier, and 3) curcumin extract.
  Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. Blood samples will be collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10 and 24h after taking the supplement. Each participant will perform all three treatments, with a minimum of 7 days between treatments. A questionnaire will document the side effects felt by participants.

SUMMARY:
Curcumin is a molecule soluble in fat. It has multiple health benefits. Indeed, it has anti-inflammatory and anti-oxidant properties. Curcumin could play a role in preventing diseases such as cancer, inflammatory, cardiovascular and neurodegenerative diseases. Omega-3 fatty acids are also important for good health, as they have positive effects on the cardiovascular and neurological systems. However, curcumin is poorly absorbed by the body when provided in supplements. In order to improve curcumin's absorption, a natural health product that combines curcumin and omega-3 fatty acids has been developped. The goal of this project is therefore to determine the absorption of curcumin when administered in combination with omega-3 fatty acids esterified in monoacylglycerol (MAG). This combination will be compared with a curcumin extract alone or in rice oil. A pharmacokinetic study will be carried out for each of the formulations. Pharmacokinetics (PK) is defined as monitoring the blood concentrations of curcumin over a 24-hour period after taking one of the three different supplements.

DETAILED DESCRIPTION:
15 men and 15 women in good health conditions will be recruited for this project. The study has a randomized double-blinded crossover design with three treatments that include an equal dosage of curcumin as follows :

* 400 mg of curcumin extract,
* 400 mg of curcumin in rice oil,
* 400 mg of curcumin extract + 1.5 g omega-3 in MAG form.

For each of the above listed products, a natural product number (NPN) was requested to Health Canada and these number are currently pending.

Each participant will consume each of the three treatments in a random order with a minimum of 7 days washout phase between both treatments. Blood samples will be collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10, and 24h (10 blood samples per participant per treatment) after taking the single dose intake. A questionnaire will allow documenting side effects throughout the study period. The analyses will be performed by ultra-high-performance liquid chromatography couples to a quadrupole mass spectrometer (UPLC/MS/MS). Samples will be analyzed in a blinded manner such that the student and research assistant will be blinded from the type of treatment and the time point they are analyzing. After performing all the analyses, sample identification will be decoded and pharmacokinetic data of the curcuminoids in each of the treatments will be plotted on a plasma concentration vs time curve. The parameters below will be calculated:

* Area under the curve (AUC) 0-24h (bioavailability);
* Area under the curve (AUC) 0-6h (absorption);
* Maximum concentration (Cmax);
* Time to reach the maximum concentration (Tmax);
* Half-life (if available).

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 50 years old (inclusive).
* Body mass index between 18,5 and 34,9 at the selection visit (inclusive).
* Normal to moderately high lipidemia (total cholesterol ≤ 240 mg / dl; LDL ≤ 160 mg / dl; Triglyceride ≤ 199 mg / dl).
* Women of child bearing potential must accept to use an effective contraceptive method for the duration of the study.

Exclusion Criteria:

* Allergy to fish or seafood.
* Special diet like a vegetarian or vegan diet.
* Tobacco.
* History of current or past alcohol and / or drug abuse.
* Current or past performance athlete.
* Malnutrition (assessed by albumin, hemoglobin and blood lipid levels).
* People consuming omega 3 fatty acid or curcumin supplements for more than 6 months.
* Medication affecting fat absorption (ie, Orlistat, Alli, etc.).
* Medication which interferes with the metabolization of the medication (ie, anticoagulants like coumadin or warfarin, aspirin is not an exclusion criterion (Watson et al, 2009))
* Medication which affects lipid metabolism (ie, all types of drugs to lower cholesterol or triglycerides).
* Medication which curcumin interacts with : angiotensin II blockers (losartan, valsartan), β-blockers (talinolol, celiprolol), calcium channels blockers (nifedipine), 3-hydroxy-3-methyl-glutaryl-coenzyme A reductase (HMG CoA) reductase inhibitors (rosuvastatin), antineoplastic agents (docetaxel, etoposide, tamoxifen, everolimus, sirolimus), antibiotics (norfloxacin), antidepressant (midazolam), sulfonamides (sulfasalazine), antidiabetics (gliclazide).
* Pregnant women or nursing women.
* Menopause or pre-menopause with amenorrhea > 6 months.
* Systemic disease: vasculitis, Lupus Erythrocyte Disseminated (SLE), sarcoidosis, cancer (except if in remission for more than 10 years and without cerebral involvement), uncompensated hypothyroidism, vitamin B12 deficiency not supplemented and / or complicated, diabetes, severe renal insufficiency.
* Abnormal liver, kidney or thyroid function; these conditions will not exclude a patient if he / she has been stabilized on treatment for at least 3 months and there has been no recent change in his / her medication.
* Cardiac event or recent major surgery (<6 months).
* History of thrombosis or haemorrhagic diathesis.
* Malabsorption disease such as pancreatitis, Crohn's disease or has had bariatric surgery.
* Neurodegenerative disease (Parkinson disease).
* Genetic disorder (Down syndrome).
* Known psychiatric history: schizophrenia, psychotic disorders, major affective disorder (bipolar disorder and major depression <5 years), panic disorder, Compulsive Obsessive Compulsive Disorder (OCD).
* Neurological disorder (Epilepsy, cerebral trauma with loss of consciousness, subarachnoid hemorrhage).
* Person who has donated blood or had significant blood loss in the 30 days prior to the start of the study.
* Not available to perform the 3 treatments.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 15 men and 15 women
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Determine the bioavailability of curcumin in combination with fish oil, rice oil or alone: Calculating the area under the curve (AUC) 0-48h as the first parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. UPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10 and 24 hours post-treatment.
  Plasma curcumin levels will be measured by ultra-performance liquid chromatography (UPLC), each sample being performed randomly blindly. After UPLC analyzes, area under the curve (AUC) 0-48 hours will be calculated, as the first parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of curcumin in combination with fish oil, rice oil or alone: Calculating the AUC 0-6h (absorption study) as the second parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. UPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10 and 24 hours post-treatment.
  Plasma curcumin levels will be measured by ultra-performance liquid chromatography (UPLC), each sample being performed randomly blindly. After UPLC analyzes, AUC 0-6 hours (absorption study) will be calculated, as the second parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of curcumin in combination with fish oil, rice oil or alone: Calculating the maximum concentration as the third parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. UPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10 and 24 hours post-treatment.
  Plasma curcumin levels will be measured by ultra-performance liquid chromatography (UPLC), each sample being performed randomly blindly. After UPLC analyzes, maximum concentration will be calculated, as the third parameter of the PK. Statistical analyzes will then be performed on this PK parameter.
Determine the bioavailability of curcumin in combination with fish oil, rice oil or alone: Calculating the time when the maximum concentration is reached, as the fourth parameter of the PK | Treatments are randomly assigned on days 1, 8 and 15 of the clinical study. UPLC analyzes will be measured on plasma from blood samples collected at time 0, 1, 2, 3, 4, 5, 6, 8, 10 and 24 hours post-treatment.
  Plasma curcumin levels will be measured by ultra-performance liquid chromatography (UPLC), each sample being performed randomly blindly. After UPLC analyzes, time when the maximum concentration is reached will be calculated, as the fourth parameter of the PK. Statistical analyzes will then be performed on this PK parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Plourde, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada